CLINICAL TRIAL: NCT02260960
Title: The Influence of PRN Dry Eye Omega-3 Nutritional Regimen on Tear Osmolarity In Cases Of Dry Eye Disease.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Physician Recommended Nutriceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRN 20142
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Omega-3 (Experimental): Reesterified Triglyceride form omega 3
  Interventions: Dietary Supplement: Omega-3 (Triglyceride form)
- Placebo (Placebo Comparator): safflower oil
  Interventions: Dietary Supplement: Omega-3 (Triglyceride form)

INTERVENTIONS:
Dietary Supplement: Omega-3 (Triglyceride form)

SUMMARY:
The investigators hypothesize that oral omega-3-acid triglyceride form will decrease dry-eye related symptoms as well as clinical markers associated with dry eye disease (TearOsmolarity, Schirmer-1 test values, corneal staining, and fluorescein tear break-up time) when compared to administration of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 90 at the time of informed consent
* Subjects experiencing dry eye based on a global clinical assessment by the attending clinician, subject complaint of dry eye symptoms
* Presence or History of Tear Osmolarity (Appendix 2) equal to or greater than 312 mOsm/L in at least one eye
* Presence or History of Meibomian Gland Dysfunction (Grade 1 or 2) in at least one eye

Exclusion Criteria:

* Allergy to fish oil or safflower oil
* Clinically significant eyelid deformity or eyelid movement disorder that is caused by conditions such as notch deformity, incomplete lid closure, entropion, ectropion, hordeola or chalazia
* Previous ocular disease leaving sequelae or requiring current topical eye therapy other than for DED, including, but not limited to: active corneal or conjunctival infection of the eye and ocular surface scarring Active ocular or nasal allergy
* LASIK or PRK surgery that was performed within one year of the Screening Visit or at any time during the study
* Ophthalmologic drop use within 2 hours of any study visits. Any OTC habitual artificial tear should be continued at the same frequency and no change in drop brand
* Contact lens wear within 12 hours of any study visits
* Pregnancy or lactation during the study
* Abnormal nasolacrimal drainage (by history)
* Punctal cauterization or punctal plug placement within 60 days of screening
* Prohibited Medications - Cyclosporine (Restasis®); any topical prescription medications (i.e., steroids, NSAIDs, etc); glaucoma medications; oral tetracyclines or topical macrolides; oral nutraceuticals (flax, black currant seed oils, etc…) within 3 weeks (21 days) of Screening and at any time during the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Tear Osmolarity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice Epitropoulos, MD, Principal Investigator — The Eye Center of Columbus
Locations (1):
- The Eye Center of Columbus, Columbus, Ohio, United States